CLINICAL TRIAL: NCT03678766
Title: Targeting Food Cue Reactivity and Satiety Sensitivity to Decrease Binge Eating and Weight
Brief Title: CHARGE: Controlling Hunger and ReGulating Eating
Acronym: CHARGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kerri Boutelle, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 181015
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Binge-Eating Disorder; Overweight; Obesity
Keywords: Overweight; Obesity; Binge Eating; Overeating; Body Mass Index; Weight; Treatment; Intervention; Behavioral Treatment
MeSH Terms: conditions — Binge-Eating Disorder; Overweight; Obesity; Bulimia; Hyperphagia; Body Weight | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regulation of Cues (ROC) (Experimental): The ROC program provides psychoeducation, coping skills, self-monitoring and experimental learning.
  Interventions: Behavioral: Regulation of Cues (ROC)
- Cognitive Behavior Therapy (CBT) (Experimental): CBT provides coping skills, self-monitoring, and goal setting.
  Interventions: Behavioral: Cognitive Behavior Therapy (CBT)

INTERVENTIONS:
Behavioral: Regulation of Cues (ROC) — Participants are provided information about basic learning theory and how physiological responses to food cues develop and can be managed. Lack of sensitivity to appetite and satiety cues and increased sensitivity to food cues will be discussed. Coping skills are presented to assist in mastery and toleration of food cue sensitivity. Participants will complete experiential learning exercises with food, and taught to monitor their hunger, satiety, and cravings. The physical activity program will focus on increasing both lifestyle activity and structured exercise programs.
  Other Names: ROC
  Arms: Regulation of Cues (ROC)
Behavioral: Cognitive Behavior Therapy (CBT) — Participants are taught to identify problems in eating, thinking, and mood patterns that served to trigger binge episodes through self-monitoring and to gradually develop alternative patterns aimed at facilitating healthy, binge-free eating patterns. Participants are taught to eat a healthy variety of foods and reducing the avoidance of "forbidden" foods that are typically consumed during a binge.
  Other Names: CBT
  Arms: Cognitive Behavior Therapy (CBT)

SUMMARY:
The objectives of this proposed study are: 1) to evaluate feasibility and acceptability of a novel intervention, Regulation of Cues (ROC), and Cognitive Behavior Therapy (CBT), and 2) to evaluate the efficacy of both treatments on reduction of binge eating and weight loss among 120 Veterans with subclinical or clinical Binge Eating Disorder (BED) with comorbid overweight/obesity (OW/OB).

DETAILED DESCRIPTION:
The investigators have developed a new model for the treatment of obesity, called Regulation of Cues (ROC), which is based on Schachter's Externality Theory. This study will compare ROC with Cognitive Behavior Therapy for individuals with Binge Eating Disorder. The investigators will recruit and randomize 120 male and female Veterans with BED and subclinical BED with comorbid overweight/obesity, provide 5 months of treatment and follow participants for 6-months post-treatment. Participants will complete assessments at baseline, mid-treatment (week 9), post-treatment (week 20), and 6-month follow-up (week 44). This study will be the first to contribute to a body of literature developing treatments for BED and overweight/obesity in the Veterans Affairs (VA) and/or military health care systems.

ELIGIBILITY:
Inclusion Criteria:

1. All participants will be Veterans between the ages of 18-65 meeting criteria for overweight, with a 45≥ BMI ≥25.
2. Participants will meet Diagnostic and Statistical Manual-5 (DSM-5) criteria for BED or subclinical BED
3. Participants will be willing and able to participate in assessment visits and treatment sessions at University of California, San Diego (UCSD).
4. Participants will be able to provide data in English through interviews and questionnaires and understand treatment materials in English.
5. Participants will be willing to maintain contact with the investigators for 11 months.
6. Participants will be free of serious or unstable medical (current symptoms of angina, stroke, heart disease or other serious medical condition that would make physical activity unsafe or impossible at a moderate level) or psychiatric illness (i.e., active suicidal ideation, history of suicide attempt within 1 year, current unmanaged psychosis, manic episode, anorexia nervosa, bulimia nervosa, or substance abuse within the past year) or psychosocial instability (e.g., homelessness) that could compromise study participation.
7. Participants will be free from conditions in which exercise or weight loss will be detrimental to the participant's health (e.g., pregnancy); pharmacotherapy for obesity or binge eating disorder (e.g., Orlistat or Meridia) or bariatric surgery within the past 6 months or planning to start such treatments in the next 11 months.
8. Participants will not be moving out of the San Diego area for the duration of their study enrollment (11 months).
9. Participants will not be pregnant, planning to get pregnant in the 11-month study period or lactating.
10. Participants will not be participating in group or individual psychotherapy for binge eating or weight management.
11. Participants with medical or psychological problems or taking medications that could make adherence with the study protocol difficult or dangerous will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Attendance | Post-Treatment (5 months following baseline)
  The number of treatment visits attended
Acceptability | Post-Treatment (5 months following baseline)
  Average likert ratings to questions, such as "How much did you enjoy the treatment?" and "How helpful did you find the treatment?"
Binge Eating as measured by the Eating Disorder Examination (EDE) | Changes from baseline at an average of 9 weeks, 20 weeks, and 44 weeks
  Diagnosis of Binge Eating Disorder (BED) and subclinical BED, number of OBEs (large amount of food and loss of control), objective overeating episodes (large amount of food without loss of control), and SBEs (lack of large amount of food with loss of control) determined by responses to the EDE.
Binge Eating as measured by the Binge Eating Scale (BES) | Changes from baseline at an average of 9 weeks, 20 weeks, and 44 weeks
  Dimensional score of binge eating consisting of items to describe binge eating behaviors and feelings and cognitions associated with binge eating.
Binge Eating as measured by the Eating Disorder Examination-Questionnaire (EDE-Q) | Changes from baseline at an average of 9 weeks, 20 weeks, and 44 weeks
  Three question items from the questionnaire to calculate the number of binge eating episodes and number of days participants experienced a binge eating episode.
Body Mass Index (BMI) as measured by weight and height | Changes from baseline at an average of 9 weeks, 20 weeks, and 44 weeks
Energy intake | Changes from baseline at an average of 20 weeks and 44 weeks
  Calorie intake estimated by 24-hour dietary recalls on 3 non-consecutive days

SECONDARY OUTCOMES:
Satiety Responsiveness | Changes from baseline at an average of 9 weeks, 20 weeks, and 44 weeks
  Self-reported satiety responsiveness measured by the Adult Eating Behavior Questionnaire (AEBQ)
Food Responsiveness | Changes from baseline at an average of 9 weeks, 20 weeks, and 44 weeks
  Self-reported food responsiveness measured by the Adult Eating Behavior Questionnaire (AEBQ)
Reward-Based Eating | Changes from baseline at an average of 9 weeks, 20 weeks, and 44 weeks
  Scales to evaluate reward-related eating measured by the Reward-Based Eating Drive Scale (RED-13)

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, Ph.D, Principal Investigator — UCSD
Locations (1):
- UCSD Center for Healthy Eating and Activity Research (CHEAR), La Jolla, California, United States

REFERENCES:
- [Background] Boutelle KN, Zucker NL, Peterson CB, Rydell SA, Cafri G, Harnack L. Two novel treatments to reduce overeating in overweight children: a randomized controlled trial. J Consult Clin Psychol. 2011 Dec;79(6):759-71. doi: 10.1037/a0025713. PMID 22122291
- [Background] Boutelle KN, Zucker N, Peterson CB, Rydell S, Carlson J, Harnack LJ. An intervention based on Schachter's externality theory for overweight children: the regulation of cues pilot. J Pediatr Psychol. 2014 May;39(4):405-17. doi: 10.1093/jpepsy/jst142. Epub 2014 Jan 23. PMID 24459240
- [Derived] Boutelle KN, Afari N, Obayashi S, Eichen DM, Strong DR, Pasquale EK, Peterson CB. Regulation of Cues vs Cognitive Behavioral Therapy for Binge Eating and Weight Loss Among Veterans: A Feasibility and Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2525064. doi: 10.1001/jamanetworkopen.2025.25064. PMID 40758351
- [Derived] Boutelle KN, Afari N, Obayashi S, Eichen DM, Strong DR, Peterson CB. Design of the CHARGE study: A randomized control trial evaluating a novel treatment for Veterans with binge eating disorder and overweight and obesity. Contemp Clin Trials. 2023 Jul;130:107234. doi: 10.1016/j.cct.2023.107234. Epub 2023 May 19. PMID 37210072